CLINICAL TRIAL: NCT03270800
Title: A Randomized, Double-blind, Adjuvant-controlled Phase 1a/b Study on Safety and Tolerability With Ascending Multiple Doses of IMX101 in H. Pylori-negative and H. Pylori-infected Healthy Volunteers
Brief Title: Phase 1a/b Study on Safety of IMX101 in H. Pylori-negative and H. Pylori-infected Healthy Volunteers
Acronym: IMX-02
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImevaX (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-004761-82
Record Dates: First submitted 2017-02-22; First posted 2017-09-01 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Helicobacter Pylori Infected Subjects; Helicobacter Pylori Naive Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMX101 vaccine as intradermal and sublingual application (Experimental): IMX101 vaccine will be administered intradermally and sublingually
  Interventions: Biological: IMX101 vaccine
- CTA control as intradermal and sublingual application (Experimental): CTA mucosal adjuvans will be administered intradermally and sublingually
  Interventions: Biological: CTA control

INTERVENTIONS:
Biological: CTA control — Sublingual and intradernal application of a mucosal adjuvance, drug product is not yet on the market.
  Arms: CTA control as intradermal and sublingual application
Biological: IMX101 vaccine — Sublingual and intradermal application of a vaccine, drug product is not yet on the market.
  Arms: IMX101 vaccine as intradermal and sublingual application

SUMMARY:
A Phase 1, multi-center, randomised, double-blind and adjuvant-controlled study to evaluate the safety, tolerability, and efficacy of IMX101 in H. pylori-negative and H. pylori-infected healthy volunteers.

The study will be conducted in 2 phases. Phase A: Study design contains 6 cohorts, each containing 8 subjects. Three cohorts (24 subjects) will be H. pylori-negative and 3 cohorts will be H. pylori-infected. Subjects fulfilling the inclusion criteria will be assigned to one of 3 sequential dose cohorts with a 3:1 randomisation to IMX101 or to CTA within each cohort.

Phase B: Two cohorts with H. pylori-infected subjects can be expanded up to 20 subjects in each cohort. The decision whether to expand the cohorts will be taken by the Sponsor and the DSMB, as soon as the results of the safety and efficacy analyses are available.

Up to 72 subjects collectively in Phases A & B will be recruited. depending on immunogenicity status.

ELIGIBILITY:
Inclusion Criteria:

* H. pylori-infected subjects: Confirmed H. pylori infection by urea breath test and serology.

H. pylori-negative subjects: Presenting no H. pylori infection by urea breath test and serology.

* Men and women aged ≥18 years and ≤ 50 years.
* Female subjects must either be of non-childbearing potential or use highly effective methods of contraception for at least 1 month prior to Screening and 1 month after end of study participation (see section pregnancy and contraceptives).
* Women with a negative serum test at Screening (V2) and women of childbearing potential additionally with a negative urine pregnancy test at each visit (except V1 and FU V10/V12).
* Have given written informed consent prior to admission to the study in accordance with ICH-GCP and local legislation.
* Ability to comply with the requirements of the study protocol.

Exclusion Criteria:

* History of successful treatment for H. pylori infection.
* Regular use (once a week or more) of diclofenac, other non-steroidal anti-inflammatory drugs (NSAIDs), e.g. acetylsalicylic acid (Aspirin®), or proton pump inhibitor (PPI). Additionally, PPI is used within 2 weeks prior to V1 and V11.
* Use of anticoagulants (i.e. heparin, coumarin derivatives, e.g. Marcumar®).
* Use of antibiotics employed in H. pylori therapy within the month prior to study entry (V1) as well as 1 month prior to each endoscopy (V3 and V9/V11).
* Recent or current (within the last 6 months) systemic corticosteroid use including inhaled corticosteroids. Topical corticosteroid medication is allowed.
* Current or previous gastric ulcer diseases or preneoplastic changes in the stomach mucosa according to medical records or endoscopy findings confirmed by histological assessment at Baseline (V3).
* Current or previous medically significant gastroduodenal disease.
* Preceding cholera immunisation or disease.
* Uncontrolled hypertension or orthostatic hypotension.
* Body mass index (BMI) ≤ 18 or ≥ 30.
* Poorly-controlled type I or type II diabetes mellitus (glycosylated haemoglobin [HbA1c] ≥ 7.5% within the last 6 weeks) and subjects requiring insulin treatment.
* History, evidence or suspicion of tumour burden.
* Epilepsy or seizure disorder.
* Bleeding diathesis.
* Positive viral serology screening result for hepatitis B surface antigen (HBS Ag), antibodies to hepatitis C virus (HCV Ab), or human immunodeficiency virus (HIV) type 1 and 2.
* Known significant allergic reaction to any drug as determined by the investigator, such as anaphylaxis requiring hospitalisation.
* A history of active alcohol abuse or drug addiction.
* Administration of a live vaccine within 90 days prior to the first study immunisation (V4) and throughout the study.
* Receipt of blood, blood products or plasma derivatives 30 days prior to study entry (V1).
* Pregnancy or lactation.
* Participation in a clinical study within 30 days prior to admission to the study if investigational or marketed drug were employed. Any disease or condition which in the Investigator's opinion would exclude the subject from the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2018-12-23 (Actual); Study Completion 2018-12-23 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of IMX101 | 215 days
  All subjects who received at least one dose of the IMP will be included in the safety analysis by following parameters:
  -Adverse events: AEs will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA). Separate analyses will be conducted using severity, seriousness, and relationship to the IMP. Treatment-emergent adverse events (TEAEs) will be summarised and tabulated according to the primary system organ class and preferred term.
  * Clinical laboratory and other safety measures Haematology and clinical chemistry will be summarised with descriptive statistics for absolute values und changes from Baseline by visit. Urine dipstick test will be summarised with frequency tables by visit.
  * Vital signs Vital signs will be summarised with descriptive statistics for absolute values und changes from Baseline by visit.
  * Local tolerability Injection site assessments will be summarised in frequency tables when the collected data allow for this.

SECONDARY OUTCOMES:
Determination of immune Responses | 215 days
  Humoral and cellular immune Response towards IMX101 and detection of inhibitory antibodies
  Secondary Endpoint(s):
  * Detection of vaccine-antigen specific antibodies by Enzyme linked immunosorbent assay (ELISA) at V6, V7, V8 and V9 in the non-infected subjects and at V6, V7, V8, V9, V10 and V11 in the H.pylori infected subjects.
  * Detection of inhibitory antibodies blocking H.pylori gGT enzymatic activity at V6, V7, V8 and V9 in the non-infected subjects and at V6, V7, V8, V9, V10 and V11 in the H.pylori-infected subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Zivotic, Principal Investigator — CTC-NORTH
Locations (2):
- Germany (2):
  - ClinicalTrial Site, Hamburg
  - Clinical Trial Site, Munich

IPD SHARING:
Plan to Share IPD: Undecided